CLINICAL TRIAL: NCT03166566
Title: Laminar Drainage Implant: Safety of a Novel Surgical Treatment for Refractory Glaucoma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, SÉRGIO JACOBOVITZ, co-advisor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAAE 0194.0.203.203.09
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma; Blindness, Acquired; End-Stage Glaucoma; Glaucoma Traumatic
Keywords: glaucoma; glaucoma surgery; glaucoma drainage device; glaucoma implant; blindness
MeSH Terms: conditions — Glaucoma; Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laminar drainage implant surgery (Other): patients included and operated
  Interventions: Device: Laminar drainage implant surgery.

INTERVENTIONS:
Device: Laminar drainage implant surgery. — A clear corneal traction suture was placed to achieve superior-temporal quadrant exposure, where a 90° conjunctival fornix-based flap was made, associated with two radial relaxing incisions. A half-thickness scleral tunnel (4.5 mm from the limbus and 4.0 mm wide) was made using a crescent blade and a superior-temporal iridectomy was performed through . Then, the tunnel end was shunted to the AC using a 1.5-mm-wide blade with a sharp tip. The LDI was inserted into the scleral tunnel so that its tip was positioned in the AC periphery and the implant was anchored to the sclera using 7-0 polypropylene thread with two separate sutures. Next, fistula function was assessed by the aqueous humor leakage test at the scleral tunnel entry site. Then, the conjunctiva was repositioned and running sutures were performed with 7-0 polyglactin for the relaxing incisions and mattress sutures were performed in the limbus using 10-0 nylon.

SUMMARY:
Purpose: To assess the feasibility of a surgical technique and present the preliminary safety results of a new glaucoma device devoid of a tube in painful blind eyes.

Methods: Fifteen end-stage glaucomatous eyes without light perception vision were treated with a novel laminar drainage implant. Intraocular pressure was measured preoperatively and up to 24 months after surgery using a Goldmann applanation tonometer. A scale ranging from 0 to 10 was used to evaluate ocular pain. Conjunctival hyperemia, discharge, erosion or retraction, aqueous humor leakage, corneal edema, hyphema, anterior chamber cells and depth, dislocation of the implant, and filtering bleb height were assessed by slit-lamp biomicroscopy. Anterior segment optical coherence tomography was also assessed.

DETAILED DESCRIPTION:
Methods: Light perception was tested in the preoperative assessment. The following parameters were evaluated at the pre- and postoperative visits: morning Goldmann applanation tonometry; anterior segment biomicroscopy, gonioscopy, and eye pain intensity. Postoperative visits occurred on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years. The criteria for IOP reduction success were 15 mmHg and a 20% reduction compared to the baseline preoperative IOP. Biomicroscopy variables included the presence or absence of hyperemia, discharge, conjunctival erosion and retraction, aqueous humor leakage (Seidel test), corneal edema, hyphema, AC reaction and depth, and device dislocation. A shallow AC was considered a Spaeth classification grade of I or II and a flat AC was considered grade III. A filtering bleb height above the LDI profile was considered elevated; otherwise, it was classified as flat. Gonioscopy was performed preoperatively and postoperatively. Ocular pain intensity was assessed before and after surgery using a verbal Numerical Rating Scale ranging from zero to 10, with zero representing the absence of pain and 10 representing the worst eye pain ever felt before surgery.

Anterior segment optical coherence tomography (AS-OCT) (Visante®, Carl Zeiss Meditec®, Inc., Dublin, CA, USA) was performed postoperatively at the highest resolution (enhanced high-resolution corneal mode).

Reoperations to unblock the internal ostium were not considered failures; thereafter, the day of the second surgery was considered postoperative day 0.

LDI A human LDI was designed by one of the authors (S.J.) after a preclinical trial in rabbits with a similar device. It is a 150-µm-thick foil made of polymethylmethacrylate (PMMA), composed of three functional areas (Fig. 1): 1) the tip, which has a triangular shape and is inserted into the AC angle; 2) the intermediate portion, which has a rectangular shape (4.5 mm long × 4.0 mm wide) and is positioned inside a scleral tunnel; and 3) the posterior plate, which has a round shape (diameter = 12.5 mm) and is positioned between the sclera and conjunctiva. The LDI plate is positioned only 4.5 mm from the corneoscleral limbus and no allograft coverage is necessary. Its hypothetical mechanism of action is similar to those of popular GDIs and shunts the aqueous humor from the AC to the subconjunctival plate. The difference between their designs is the absence of a tube in the LDI. Thus, aqueous humor drainage is supposed to occur in the space between the inner walls of the scleral tunnel and LDI and/or thought is cleft.

LDI Surgery All surgeries were performed under local peribulbar anesthesia by the same surgeon (S.J.).

Statistical Analysis The sample size was calculated based on IOP standard deviation values from the first seven patients who were operated on (an internal pilot study) while considering 15 mmHg as the minimal clinically relevant difference to be detected.

Histogram inspection and Shapiro-Wilk tests were used to assess the assumption of the normality of variables. Wilcoxon's rank-sum test was used to compare the median pain intensity at each postoperative visit to that at the preoperative visit. Conjunctival hyperemia, AC cells, corneal edema, and hyphema variables were analyzed using McNemar's test. The comparison between the pre- and postoperative mean IOP was performed using Student's two-tailed paired t-test. Results were analyzed using SPSS® (Statistical Package for the Social Sciences) for Windows version 18.0 (IBM, Chicago, IL, USA) and the alpha level (type I error) was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older with a painful blind eye refractory to clinical treatment and an intraocular pressure (IOP) ≥ 30 mmHg.

Exclusion Criteria:

* eyes with extensive conjunctival scarring, a disorganized anterior segment, or retinal detachment identified by ophthalmoscopy or B-scan ultrasonography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
Change for baseline of intra-ocular pressure (Goldmann applanation tonometry) | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  The criteria for IOP reduction success were 15 mmHg and a 20% reduction compared to the baseline preoperative IOP.

SECONDARY OUTCOMES:
Ocular pain intensity ratting change from baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  Ocular pain intensity was assessed before and after surgery using a verbal Numerical scale.
Conjunctival discharge presence/absence change from baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  conjunctival discharge was assessed by slit-lamp examination
Conjunctival erosion or retraction appearence after surgery | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  Presence or abscence of conjunctival tissue erosion or retraction, caused by the tested
Corneal edema presence change from baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  assessed by slit-lamp biomicroscopy was classified as "present" or "abscent"
Anterior chamber depth (gonioscopy) change from baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  A shallow AC was considered a Spaeth classification grade of I or II and a flat AC was considered grade III. A filtering bleb height above the LDI profile was considered elevated; otherwise, it was classified as flat
Optic coherence tomography (OCT) assessment qualitative study after surgery | from 6 months to two years after surgery.
  OCT image were obtained in 8 patients after surgery in order to imaging study the implant and its relation with the eye structures.
Filtering bleg height variation from baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  bleb heigh(if not above implant profile)t was slit-lamp assessed. classified as "elevated" (above implant profile) or "flat"
Conjunctival hyperemia change comparing to baseline | on days 1, 3, 7, 14, and 30, once a month up to 6 months, and every 6 months from 6 months to 2 years.
  conjunctival inflamation graduation assessed by slit-lamp examination ("present or abscent")

CONTACTS AND LOCATIONS:
Overall Officials: Sebastião C. Sobrinho, Md, Ph.D, Principal Investigator — Hospital São Geraldo-Universidade Federal de Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolf A, Hod Y, Buckman G, Stein N, Geyer O. Use of Autologous Scleral Graft in Ahmed Glaucoma Valve Surgery. J Glaucoma. 2016 Apr;25(4):365-70. doi: 10.1097/IJG.0000000000000232. PMID 25719229
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Result] Christakis PG, Zhang D, Budenz DL, Barton K, Tsai JC, Ahmed IIK; ABC-AVB Study Groups. Five-Year Pooled Data Analysis of the Ahmed Baerveldt Comparison Study and the Ahmed Versus Baerveldt Study. Am J Ophthalmol. 2017 Apr;176:118-126. doi: 10.1016/j.ajo.2017.01.003. Epub 2017 Jan 17. PMID 28104418
- [Result] Thieme H, Choritz L, Schuart C, Wecke T. [Tube versus trabeculectomy study]. Ophthalmologe. 2013 Aug;110(8):728-32. doi: 10.1007/s00347-013-2840-z. German. PMID 23873397
- [Result] Aref AA, Gedde SJ, Budenz DL. Glaucoma Drainage Implant Surgery. Dev Ophthalmol. 2017;59:43-52. doi: 10.1159/000458485. Epub 2017 Apr 25. PMID 28442686